CLINICAL TRIAL: NCT05048966
Title: Comparison of Two Group Wellness Interventions for Individuals With Neurologic Conditions and Their Support Persons: A Randomized Clinical Trial
Brief Title: Comparison of Two Group Wellness Interventions for Individuals With Neurologic Conditions and Their Support Persons
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: University of Michigan (Other); Franciscan Health (Unknown); Rehabilitation Hospital of Indiana (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Denise Krch, Senior Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-1157-21
Record Dates: First submitted 2021-08-26; First posted 2021-09-17 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Traumatic Brain Injury; Mild Traumatic Brain Injury; Alzheimer's Disease; Brain Injury Traumatic Moderate; Brain Injury Traumatic Severe; Dementia
Keywords: Traumatic Brain Injury; Mild Traumatic Brain Injury; Alzheimer's Disease; Caregivers; Moderate Traumatic Brain Injury; Severe Traumatic Brain Injury; Alzheimer's disease related dementia; Support Persons
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Wellness Class 1 (Experimental)
  Interventions: Behavioral: Group Wellness Class 1
- Group Wellness Class 2 (Active Comparator)
  Interventions: Behavioral: Group Wellness Class 2

INTERVENTIONS:
Behavioral: Group Wellness Class 1 — Twelve weekly online group wellness sessions for individuals with the disability and their support person. Each class will last for approximately 2 hours.
  Arms: Group Wellness Class 1
Behavioral: Group Wellness Class 2 — Twelve weekly online group wellness sessions for individuals with the disability and their support person. Each class will last for approximately 2 hours.
  Arms: Group Wellness Class 2

SUMMARY:
Approximately 5.3 million people live with a long-term disability resulting from a traumatic brain injury (TBI) and between 5-8% of those older than 60 suffer from Alzheimer's disease or other forms of dementia (ADRD). Consequences of these conditions can result in dramatic and persistent changes in functioning, impacting not only the patients, but also loved ones who become informal support persons. Many existing services help the family in the moment, but do not address long-term wellness. Thus, the purpose of this research study is to compare the effect of two different types of group wellness treatments for individuals with chronic mild TBI, moderate to severe TBI, and ADRD and their support persons.

DETAILED DESCRIPTION:
The study will involve three sites, with a different clinical population targeted at each site. Kessler Foundation will serve as the Coordinating Center and will enroll individuals with moderate/severe TBI. Franciscan Health in Indiana and University of Michigan will serve as partnering sites and will enroll individuals with chronic mild TBI and ADRD respectively. The research protocols at each site will be unique to the patient population, but harmonized through unified project goals: 1) to evaluate the efficacy of two different online group wellness treatments designed to improve self-efficacy and quality of life, and 2) to determine whether patient neurobehavioral functioning moderates the relationship between treatment outcomes and burden in caregivers, and 3) to determine the neural, behavioral, and blood biomarkers that best predict treatment efficacy. It is expected that findings generated from this study will lead to improved holistic approaches for brain injury and dementia systems of care.

ELIGIBILITY:
For individuals with moderate/severe TBI:

Inclusion Criteria:

* age 18-64
* at least one year post injury
* can read and speak English fluently
* has a support person who is willing to participate in the study

Exclusion Criteria:

* has had a prior stroke or neurological disease other than TBI
* has unstable or uncontrolled seizures
* has been hospitalized due to a significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) in the past three months
* current alcohol and/or drug use that interferes with ability to carry out common everyday functions

For individuals with chronic mild TBI:

Inclusion Criteria:

* age 18-64
* at least 3 months post-injury
* can read and speak English fluently
* has a support person who is willing to participate in the study

Exclusion Criteria:

* has had a prior stroke or neurological disease other than mild TBI
* has unstable or uncontrolled seizures
* has been hospitalized due to a significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) in the past three months
* current alcohol and/or drug use that interferes with ability to carry out common everyday functions

For Individuals with Alzheimer's Disease Related Dementias (ADRD)

Inclusion Criteria:

* age 65 and older
* at least one-year post-diagnosis
* can read and speak English fluently
* has a support person who is willing to participate in this study

Exclusion Criteria:

* has had a prior stroke or neurological disease other than ADRD
* has unstable or uncontrolled seizures
* has been hospitalized due to a significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) in the past three months
* current alcohol and/or drug use that interferes with ability to carry out common everyday functions

For Support Persons:

Inclusion Criteria:

* is the support person of an individual with moderate/severe TBI, chronic mild TBI or ADRD who is willing to participate in the study
* can read and speak English fluently

Exclusion Criteria:

* has a significant neurological history (e.g. stroke or multiple sclerosis)
* has unstable or uncontrolled seizures
* has been hospitalized due to a significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) in the past three months
* current alcohol and/or drug use that interferes with ability to carry out common everyday functions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change on Self-Efficacy Questionnaire (SEQ) | 12 weeks (between pre- and post-testing) and 6 months (between post-testing and 6 month follow-up)
  self-report instrument that assesses an individual's and support person's self-efficacy as it relates to their ability to manage the effects of the neurologic conditions on their daily functioning
Change on Satisfaction with Life Scale (SWLS) | 12 weeks (between pre- and post-testing) and 6 months (between post-testing and 6 month follow-up)
  self-report measure that examines life satisfaction component of subjective well-being and quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States